CLINICAL TRIAL: NCT03770468
Title: Molecular Genetic, Host-derived and Clinical Determinants of Long-term Survival in Glioblastoma
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1419-BTG
Record Dates: First submitted 2018-11-18; First posted 2018-12-10 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood drawl

SUMMARY:
This pro - and retrospective multicenter clinical epidemiological study studies the molecular genetic, host-derived and clinical determinants of glioblastoma patients with an overall survival of more than 5 years. The different research focusses are:

* Identification of clinical parameters and patient characteristics / host-related factors in long-term survivors (Focus 1)
* Identification of molecular tumor characteristics in long-term survivors (Focus 2)
* Assessment of therapy-related parameters, including neuro-toxicity (Focus 3)
* Immunological studies (Focus 4)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at diagnosis
* Histopathological diagnosis of glioblastoma (reference histology available) and
* Survival >5 years from diagnosis
* Availability of tumor tissue from initial glioblastoma diagnosis (FFPE or fresh-frozen) to validate the diagnosis centrally.
* Signed consent form (living patients) or ethics approval for anonymous data collection in case of retrospective analysis of deceased patients

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioblastoma patients with overall survival > 5 years
Sampling Method: Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2015-07-05 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year from last patient in
Molecular profiling on FFPE samples | 1 year from last patient in
  Profiling for cytosine-phosphate-guanosine (CpG) methylation patterns using the Illumina 850k bead array platform
Molecular profiling on frozen samples | 1 year from last patient in
  Samples will be subjected to whole exome sequencing
Molecular profiling on frozen samples | 1 year from last patient in
  Samples will be subjected to messenger ribonucleic acid (mRNA) sequencing
Molecular profiling on frozen samples | 1 year from last patient in
  Samples will be subjected to miRNA sequencing
Molecular profiling on frozen samples | 1 year from last patient in
  Samples will be subjected to microarray-based expression profiling
Proteome profiling | 1 year from last patient in
  Tumor cells will be microdissected from frozen sections and prepared for high-resolution mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Principal Investigator — EORTC Study Coordinator
Locations (27):
- Dana-Farber Cancer Institute & Harvard Medical School, Boston, Massachusetts, United States
- Universitaetsklinikum Wien - AKH uniklinieken, Vienna, Austria
- Hopitaux Universitaires Bordet-Erasme, Brussels, Belgium
- France (8):
  - CHU Lyon - Hopital neurologique Pierre Wertheimer, Bron
  - CHRU de Lille, Lille
  - Hopitaux de Marseille - Hôpital de La Timone (APHM), Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - CHU de Nice - Hopital Pasteur, Nice
  - Hopitaux de Paris - Hopital Saint-Louis, Paris
  - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - CHU d'Amiens - CHU Amiens - Hopital Sud, Salouël
- Germany (9):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum - Essen, Essen
  - Ronellenfitsch Michael, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - UniversitaetsKlinikum Heidelberg, Heidelberg
  - Ludwig-Maximilians-Universitaet Muenchen - Campus Grosshadern, München
  - Technische Universitaet Muenchen - Klinikum Rechts Der Isar, München
  - Universitaetsklinikum Regensburg, Regensburg
- Hygeia Hospital, Athens, Greece
- Italy (2):
  - Azienda Ospedaliera Di Padova - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale San Giovanni, Torino
- Netherlands (2):
  - Amsterdam UMC - locatie VUmc, Amsterdam
  - Erasmus MC, Rotterdam
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - Univ. Spital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided